CLINICAL TRIAL: NCT06204484
Title: The Effectiveness of Deferred Adjuvant Therapy Guided by Dynamic Monitoring Minimal Residue Disease in Resectable High-risk Stage II and Low-risk Stage III Colon Cancer: an Open-label, Multicenter, Phase II Clinical Study
Brief Title: MRD-guided Deferred Adjuvant Therapy in Resectable Early-stage Colon Cancer
Acronym: MIRROR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: Guangzhou Burning Rock Dx Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Gong Chen, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MIRROR
Record Dates: First submitted 2023-11-28; First posted 2024-01-12 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Colorectal Cancer
Keywords: circulating tumor DNA; adjuvant therapy
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- MRD-negative standard adjuvant therapy (Active Comparator): In MRD-negative standard therapy groups, patients will receive 3-month capecitabine and oxaliplatin (CAPEOX) therapy.
  Interventions: Other: CAPEOX adjuvant therapy
- MRD-negative deferred adjuvant therapy (Experimental): In MRD- deferred adjuvant therapy group, patients won't get the standard CAPEOX adjuvant therapy at first. When MRD negative status turns to positive status, the 3-month CAPEOX therapy will be arranged.
  Interventions: Other: deferred CAPEOX adjuvant therapy
- MRD-positive standard adjuvant therapy (Active Comparator): In MRD-positive standard therapy groups, patients will receive 3-month CAPEOX therapy, regardless of the MRD status.
  Interventions: Other: CAPEOX adjuvant therapy
- MRD-positive intensive adjuvant therapy (Experimental): In the MRD+ intensive standard therapy group, which represents a high risk of recurrence, patients will receive 3-month modified folinic acid, fluorouracil, oxaliplatin and irinotecan (mFOLFOXIRI) intensive therapy, instead of the CAPEOX standard adjuvant therapy.
  Interventions: Other: mFOLFOXIRI intensive adjuvant therapy

INTERVENTIONS:
Other: CAPEOX adjuvant therapy — In MRD-/+ standard therapy groups, patients will receive 3-month CAPEOX therapy, regardless of the MRD status.
  Arms: MRD-negative standard adjuvant therapy; MRD-positive standard adjuvant therapy
Other: deferred CAPEOX adjuvant therapy — In MRD-negative deferred adjuvant therapy group, patients won't get the standard CAPEOX adjuvant therapy at first. When MRD negative status turns to positive status, the 3-month CAPEOX therapy will be arranged.
  Arms: MRD-negative deferred adjuvant therapy
Other: mFOLFOXIRI intensive adjuvant therapy — In the MRD+ intensive standard therapy group, which represents a high risk of recurrence, patients will receive 3-month mFOLFOXIRI intensive therapy, instead of the CAPEOX standard adjuvant therapy.
  Arms: MRD-positive intensive adjuvant therapy

SUMMARY:
The aim of this clinical trial is to test whether minimal residual disease (MRD) status detected by circulating tumor DNA (ctDNA) could be used to guide precision therapy of post-surgery in colon cancer. The colon cancers are intended for resectable colon cancer of high-risk stage II and low-risk stage III status. The main questions it aims to answer are:

1. Whether patients with MRD negative status could benefit from deferred adjuvant therapy.
2. Whether patients with MRD positive status need intensive adjuvant therapy. The qualified participants will go through two different randomized groups according to the post-surgery 1-month MRD status. In MRD negative groups, participants will be divided into standard adjuvant therapy groups and deferred adjuvant therapy groups at 1:2 ratios. In MRD positive groups, participants will be divided into standard adjuvant therapy groups and intensive adjuvant therapy groups at 1:2 ratios. All the patients will receive MRD detection every 3 months and radiological evaluation every 6 months up to 3 years, and survival follow-up up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

Participants must fit all of the following inclusion criteria to be enrolled in this study:

1. Over 18 years old (including 18 years old) and under 70 years old (including 70 years old) when signing the informed consent form;
2. The Eastern Cooperative Oncology Group (ECOG) physical status scores are 0-1 and do not deteriorate within 2 weeks before enrollment. The expected survival time is no less than 12 weeks;
3. Histological or cytological confirmed stage II high-risk and stage III low-risk none high microsatellite instability (MSI-H) colon adenocarcinoma according to the Union for International Cancer Control/American Joint Committee on Cancer (UICC/AJCC) primary tumor, regional nodes, metastasis (TNM) stage (8th edition). High-risk factors for stage II patients include: T4, poorly differentiated histology (high-grade, excluding MSI-H status), vascular invasion, neural invasion, intestinal obstruction or tumor site perforation pre-operation, positive or unknown margins, insufficient margin distance and examined lymph nodes less than 12; Stage III low-risk patients include patients with T1-3 N1 (excluding T4 or N2).
4. No evidence of distant metastasis (distant organ and/or distant lymph node metastasis) confirmed by comprehensive examination;
5. The distal end of the tumor is ≥12cm from the anal edge evaluated by pre-operative endoscopy. If the endoscopy is absent before surgery, the distance could be evaluated by radiology or during the surgery;
6. Patients who have not received neoadjuvant therapy and can achieve R0 radical resection;
7. Sufficient surgical fresh tissue samples for customized personalized MRD testing panels detected by whole exome sequencing (WES); available for preoperative blood, post-operative day (POD) 3-7 blood, and POD 21-30 blood samples for MRD testing;
8. Females of the childbearing period should take appropriate contraceptive measures and should not breastfeed from the screening stage to 3 months post-treatment. Before starting treatment, a negative pregnancy test, or one of the following criteria should be confirmed for no risk of pregnancy:

   1. Post-menopause, defined as age greater than 50 years and amenorrhea for at least 12 months after cessation of all exogenous hormone replacement therapy.
   2. Women younger than 50 years who have been amenorrhea for 12 months or more after cessation of all exogenous hormone therapy and whose luteinizing hormone (LH) and follicle-stimulating hormone (FSH) levels are within laboratory postmenopausal reference values can also be considered as post-menopausal.
   3. Have undergone irreversible sterilization surgery, including hysterectomy, bilateral oophorectomy, or bilateral salpingectomy, except bilateral tubal ligation.
9. Male participants should use barrier contraception (i.e., condoms) from the screening stage to 3 months post-treatment;
10. The participants volunteer to join in the study and signed the informed consent in writing;
11. Patients who are suitable for CAPEOX and mFOLFOXIRI adjuvant therapy.

Exclusion Criteria:

Participants who meet any of the following criteria are not eligible for this study:

1. Received any of the following treatments:

   1. Received neoadjuvant therapy in the past;
   2. Previously received any systemic chemotherapy or immunotherapy for colon cancer;
   3. Previously received any radiotherapy for colon cancer;
   4. Undergone colon cancer surgery in the past;
2. Previously or concomitantly diagnosed of other malignant tumors (except for adequately treated cervical carcinoma in situ, basal or squamous cell skin cancer);
3. Patients with other histological types rather than adenocarcinoma (such as neuroendocrine carcinoma, sarcoma, lymphoma, squamous cell carcinoma, etc.);
4. MSI-H/deficient mismatch repair (dMMR) patients;
5. Pathological, clinical, or radiologic evidence of metastatic lesions, including isolated, distant, or discontinuous intra-abdominal metastases;
6. Patients with multiple primary colorectal cancer;
7. Received other parts of open surgery rather than the colon within 14 days prior to the patient's enrollment;
8. Cannot provide surgical tissues for customized personalized MRD testing or fail to customize personalized MRD testing panels.
9. Cannot provide pre-operative blood, POD 3-7 blood, and POD 21-30 for MRD testing.
10. Suffer from other serious diseases that may affect the follow-up and short-term survival according to the judgment of the investigators;
11. Any other medical conditions and social/psychological problems, which make the patient unfit to participate in this study;
12. History of blood transfusion within 2 weeks before surgery or during surgery;
13. Those who cannot afford contrast-enhanced magnetic resonance imaging (MRI) or contrast-enhanced computed tomography (CT) for clinical follow-up;
14. Previously used Chinese patent medicine (CPM) with anti-tumor effect. Those who have used CPM with anti-tumor effect for less than 7 days, and have stopped for over 2 weeks can be enrolled in the study;
15. Have serious or uncontrolled systemic diseases (such as severe mental disease, neurological disease, epilepsy or dementia, unstable or uncompensated respiratory, cardiovascular, hepatic or renal diseases, left ventricular ejection fraction (LVEF) < 50%, evidence of uncontrolled hypertension [greater than or equal to CTCAE grade 3 hypertension despite drug therapy]); patients with dysphagia, active gastrointestinal disease, or other diseases that significantly affect drug absorption, distribution, metabolism, and excretion. Those who have ever undergone major gastrectomy;
16. Fever and body temperature above 38°C within the past 1 week, or active infection with clinical significance. Active tuberculosis. Active fungal, bacterial, and/or viral infections requiring systemic treatment;
17. Those with active bleeding or new thrombotic disease who are taking therapeutic anticoagulant drugs or have bleeding tendency;
18. Those with severe clinical abnormalities in rhythm, conduction, or morphology on the resting electrocardiogram, such as complete left bundle branch block, second-degree cardiac block, clinically significant ventricular arrhythmia, or atrial fibrillation, unstable angina, congestive heart failure, chronic heart failure with New York Heart Association (NYHA) class ≥ 2;
19. Myocardial infarction, coronary/peripheral artery bypass, or cerebrovascular accident occurred within 3 months;
20. QT interval (QTc) ≥450ms for males and ≥470ms for females in 12-lead electrocardiogram;
21. Presence of risk factors leading to prolongation of the QTc or arrhythmia, such as heart failure, ≥CTCAE (version 4.03) 2nd-degree hypokalemia (2nd-degree hypokalemia is defined as serum potassium < the lower limit -3.0mmol/L, with symptoms need treatment), congenital long QT syndrome, family history of long QT syndrome;
22. Intake of any drug known to prolong the QT interval within 2 weeks before enrollment;
23. Insufficiency of bone marrow reserve or organ function, reaching any of the following laboratory limits (without corrective treatment within 1 week before blood draw for laboratory examination):

    1. Absolute neutrophil count <1.5×109/L;
    2. Platelet count <90×109/L;
    3. Hemoglobin <90 g/L (<9 g/dL);
    4. Alanine aminotransferase >3 times the upper limit of normal (ULN);
    5. Aspartate aminotransferase>3×ULN
    6. Total bilirubin > 1.5×ULN;
    7. Creatinine > 1.5×ULN or creatinine clearance rate < 45 mL/min (calculated by Cockcroft-Gault formula);
    8. Serum albumin (ALB) <28 g/L;
24. Female subjects who are pregnant, lactating, or planning pregnancy during the study;
25. Other circumstances in which the researchers assess that participants are not fit for this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 349 (Estimated)
Dates: Start 2023-07-26 (Actual); Primary Completion 2028-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Relapse-free survival (RFS) time in MRD-negative groups | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 3 years.
  To evaluate the 3-year RFS time in MRD guided deferred adjuvant therapy groups

SECONDARY OUTCOMES:
Overall survival (OS) time in MRD-negative groups | From the date of randomization until the date of death from any cause, assessed up to 5 years.
  To evaluate the 5-year OS time in MRD-guided deferred adjuvant therapy groups
RFS time in MRD-positive groups | From the date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 3 years.
  To evaluate the 3-year RFS time in MRD-guided intensive adjuvant therapy groups
OS time in MRD+ groups | From the date of randomization until the date of death from any cause, assessed up to 5 years.
  To evaluate the 5-year OS time in MRD-guided deferred adjuvant therapy groups

OTHER OUTCOMES:
Dynamic change of MRD status and ctDNA concentration during follow-up | Assessed up to 5 years.
  The number of patients with MRD status who were consistently positive, consistently negative, and from positive to negative or from negative to positive during follow-up.
  The number of patients who had increased/unchanged ctDNA concentration or decreased ctDNA concentration.
Association between dynamic change of MRD status and ctDNA concentration and disease-free survival | Assessed up to 5 years.
  Difference in disease-free survival between patients who were consistently positive, consistently negative, and from positive to negative or from negative to positive during follow-up.
  Difference in disease-free survival between patients with increased/unchanged ctDNA concentration and decreased ctDNA concentration.
Performance of landmark MRD status and longitudinal MRD status in prediction of recurrence. | Assessed up to 5 years.
  Sensitivity, specificity, positive predictive value and negative predictive value of landmark MRD status and longitudinal MRD status in prediction of recurrence.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No